CLINICAL TRIAL: NCT03243487
Title: ThErapy Adherence Management in Veterans: A Randomized Trial
Brief Title: ThErapy Adherence Management in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Philips Respironics (Industry); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201701153; ST-17043-VAPAM-JP (Other: University of Florida Internal ID)
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Sleep Apnea of Adult
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: After undergoing screening and enrollment, participants will be assigned to either standard care follow-up or to the patient adherence monitoring service (PAMS).
Who Masked: Outcomes Assessor
Masking Description: Study participants and study staff cannot be blinded to the treatment arm to which they are randomized. Data analysis will be blinded and conducted without revealing the treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAMS service (Experimental): Study participants will be randomly assigned to have their Continuous positive airway pressure therapy (CPAP) or Bilevel Positive Airway Pressure (BiPAP) therapy followed by a structured patient adherence management service (PAMS).
  Interventions: Call to patient by sleep coach on days 3,7,14,32,45, 60, and 75 after participants begin PAP treatment. At each time frame sleep coach reviews CPAP adherence data on EncoreAnywhere (EA) a cloud based program collecting adherence data via wireless modem on CPAP units. Calls will not be made at days 7 and 14 if adherence is good. If problems are identified and cannot be handled over the telephone the problems will be escalated to VA MD or CPAP respiratory therapy (RT) providers for direct intervention. All patients are seen in sleep clinic by a VA MD sleep provider 3 months after starting treatment.
  Interventions: Behavioral: structured adherence management program
- Standard Care (SCP) (Active Comparator): Study participants will be randomly assigned to have their CPAP or BiPAP therapy followed by the current Sleep Center standard care process. This includes a telephone number that patients can call or problems and review of adherence data on EncoreAnywhere (EA) at 4 to 6 weeks after starting treatment. Patients are seen in sleep clinic by a VA MD sleep provider 3 months after starting treatment.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: structured adherence management program — Structured adherence management service (PAMS) program and a web-based information program designed for participants beginning positive airway pressure therapy
  Arms: PAMS service
Behavioral: Standard of care — Standard care provided at a VA Sleep Center for participants beginning positive airway pressure therapy
  Arms: Standard Care (SCP)

SUMMARY:
The study is a prospective, randomized, controlled trial studying adherence to positive airway pressure therapy in a population referred to the VA system for the treatment of sleep disordered breathing. The primary aim of the study is to determine if, compared to standard care provided at a VA Sleep Center, the deployment of a structured adherence management program and a web-based information program designed for participants beginning positive airway pressure therapy results in a greater portion of participants meeting Centers for Medicare & Medicaid Services (CMS) adherence requirements (use > 4 hours for >= 70% of days) at 90 days.

DETAILED DESCRIPTION:
The primary aim of the study is to determine if, compared to standard care provided at a VA Sleep Center, the deployment of a structured adherence management program and a web-based information program designed for participants beginning positive airway pressure therapy results in a greater portion of participants meeting CMS adherence requirements (use > 4hrs on >=70% of nights) at 90 days.

Secondary aims:

1. Results in higher nightly use of therapy (hours per night and % of nights with at least 4 hours of use) at 90 days
2. Results in participant satisfaction that is superior to current standard care
3. Offers operational efficiencies or economic benefits to the health care facility (reduced staff time (sleep clinic and physician), equipment consumption, unplanned participant contacts or visits, and reduced overtime)
4. Results in indirect benefits to participants (fewer clinic visits, less travel or in-clinic/ office visit waiting time)

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 to 85
* Diagnostic Apnoea-Hypopnoea Index (AHI) ≥ 15 determined by in lab polysomnography (PSG) or home sleep testing (HST) or by a sleep therapy device
* Eligible for treatment with Automatically adjusted CPAP or Automatically adjusted BiPAP
* Currently has a Smart Phone or home access (computer with internet access) to the internet based version of the software application

Exclusion Criteria:

* Participation in another interventional research concerned with sleep disorders within the last 30 days
* Major uncontrolled medical condition that would interfere with the demands of the study, adherence to PAP, or the ability to commit to follow-up assessment including conditions such as poorly managed or controlled or advanced stages of pulmonary disease, cardiac disease, neurological disease, neuromuscular disease, cancer, and renal disease.
* Prior PAP use within the previous 12 months.
* Predominantly Central Apneas (≥ 50% central apneas) or Cheyne Stokes Respiration (CSR) (≥ 20% of Total Sleep Time (TST) with CSR)
* Chronic respiratory failure or insufficiency with suspected or known neuromuscular disease, moderate chronic obstructive pulmonary disease (COPD), or any condition with an elevation of arterial carbon dioxide levels while awake or the requirement for supplemental oxygen (at night or continuous) or mechanical ventilation.
* Surgery involving the upper airway, nose, sinus, eye, teeth, or middle ear within the previous 90 days
* PAP therapy is otherwise medically complicated or contraindicated such as those with a difficult to size or adjust interface (mask) resulting in facial pain, skin irritation or trauma, or excessive air leaks

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Increase on CMS adherence requirements | at 90 days
  The requirements are greater than 4 hours use for 70% of nights

SECONDARY OUTCOMES:
Nightly use of therapy | at 90 days
  Hours per night and % of nights with at least 4 hours of use
Participant satisfaction | at 90 days
  Participants will complete at "Patients Satisfaction Survey" containing 5 questions about their satisfaction with CPAP treatment and the process of starting CPAP. There is a 5 point scale from very unsatisfied (1), unsatisfied (2), neutral (3), satisfied (4), very unsatisfied (5). Score can vary from 5 to 25. 30,
Operational efficiencies and economic benefits to the health care facility | at 90 days
  Reduced staff time (sleep clinic and physician) as evidenced by, unplanned participant contacts or visits over time

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Berry, MD, Principal Investigator — Malcom Randall VAMC
Locations (2):
- United States (2):
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antic NA, Buchan C, Esterman A, Hensley M, Naughton MT, Rowland S, Williamson B, Windler S, Eckermann S, McEvoy RD. A randomized controlled trial of nurse-led care for symptomatic moderate-severe obstructive sleep apnea. Am J Respir Crit Care Med. 2009 Mar 15;179(6):501-8. doi: 10.1164/rccm.200810-1558OC. Epub 2009 Jan 8. PMID 19136368
- [Background] Sparrow D, Aloia M, Demolles DA, Gottlieb DJ. A telemedicine intervention to improve adherence to continuous positive airway pressure: a randomised controlled trial. Thorax. 2010 Dec;65(12):1061-6. doi: 10.1136/thx.2009.133215. Epub 2010 Sep 29. PMID 20880872
- [Background] Fox N, Hirsch-Allen AJ, Goodfellow E, Wenner J, Fleetham J, Ryan CF, Kwiatkowska M, Ayas NT. The impact of a telemedicine monitoring system on positive airway pressure adherence in patients with obstructive sleep apnea: a randomized controlled trial. Sleep. 2012 Apr 1;35(4):477-81. doi: 10.5665/sleep.1728. PMID 22467985
- [Background] Aloia MS, Arnedt JT, Strand M, Millman RP, Borrelli B. Motivational enhancement to improve adherence to positive airway pressure in patients with obstructive sleep apnea: a randomized controlled trial. Sleep. 2013 Nov 1;36(11):1655-62. doi: 10.5665/sleep.3120. PMID 24179298
- [Result] Parthasarathy S, Wendel C, Haynes PL, Atwood C, Kuna S. A pilot study of CPAP adherence promotion by peer buddies with sleep apnea. J Clin Sleep Med. 2013 Jun 15;9(6):543-50. doi: 10.5664/jcsm.2744. PMID 23772186
- [Derived] Berry RB, Beck E, Jasko JG. Effect of cloud-based sleep coaches on positive airway pressure adherence. J Clin Sleep Med. 2020 Apr 15;16(4):553-562. doi: 10.5664/jcsm.8276. PMID 32022679